CLINICAL TRIAL: NCT06031753
Title: Time-restricted Eating as a Novel Approach to PCOS Remission, Compared to Guideline's Standard Hormonal Treatment.
Brief Title: Effects of Intermittent Fasting on Polycystic Ovary Syndrome (PCOS) Compared to Standard Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Superior de Investigación en Estética Médica, Nutrición y Anti-Envejecimiento (Other)
Collaborators: Centro Medico ABC (Other)
Responsible Party: Principal Investigator, Isabela von Damm Longoria, Principal investigator, Instituto Superior de Investigación en Estética Médica, Nutrición y Anti-Envejecimiento
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AYUSOP22
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Polycystic Ovary Syndrome; Insulin Resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: group 1: time restricted eating with NO hormonal treatment group 2: time restricted eating with hormonal treatment group 3: hormonal treatment with NO time restricted eating
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TRE (Experimental): Only time restricted eating was carried on by this arm, having the first meal of the day at 12:00hrs and last meal of the day at 18:00hrs. No other medication was allowed during the study for this group.
  Interventions: Behavioral: Time restricted eating
- TRE-HT (Experimental): They carried on Time Restricted eating, in combination with the oral contraceptives used for the standard hormonal treatment. First meal of the day at 12:00hrs and last meal of the day at 18:00hrs. Other than oral contraceptives, no medication was allowed during the 3 months of the study.
  Interventions: Behavioral: Time restricted eating
- HT (No Intervention): No time restricted eating was practiced by this group, only oral contraceptives were taken, serving as the control group by having the standard hormonal treatment. No modification to their daily habits and routine was made.

INTERVENTIONS:
Behavioral: Time restricted eating — Only eating windows were determined to an 6 hour period, starting at 12:00hrs and ending at 18:00hrs. After that, patients in group 1 and 2 were indicated not to consume any calories. The composition of their diet was not modified, it was assessed by performing a 24-hour recall to make sure there were no significant changes in diet composition throughout the study.
  Other Names: time restricted eating with hormonal treatment
  Arms: TRE; TRE-HT

SUMMARY:
The purpose of this study is to assess the effects of Time restricted eating in patients diagnosed with polycystic ovary syndrome, comparing it to the standard hormonal treatment.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients were given a written informed consent. Patients were recruited through social media and digital questionnaires, to make sure they met the criteria. There was a semi aleatory distribution of the patients into three different groups, one group underwent time restricted eating with no hormonal treatment (TRE group), the second group received hormonal treatment combined with time restricted eating (combined group) and the last group received only hormonal treatment (HT). PCOS was diagnosed using Rotterdam criteria, which were evaluated according to the ultrasound, blood samples and self reported menstrual cycle.

Blood samples and transvaginal ultrasound were taken at day 0 and 90 to evaluate hormonal status, including insulin and glucose.

Homeostatic assessment for insulin resistance (HOMA-IR) was calculated to determine insulin resistance, as well as metabolic disfunction.

After data collection, statistical analyses was done to determine the effect of the different approaches.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20 - 35 years
* Mild to moderate exercise at least 4 times per week
* Body Mass Index (BMI) of 20-24.9
* Diagnosis of PCOS by Rotterdam criteria
* Type of oral contraceptives: combined (estrogens and progestins) in group 1 and 2.
* PCOS Phenotype A, B, C
* nulliparity
* Signed informed consent letter

Exclusion Criteria:

* Menopause or perimenopause
* Night work shifts
* Phenotype D (without hyperandrogenism)
* Associated pathologies such as diabetes mellitus, arterial hypertension, metabolic syndrome, neoplasms, autoimmune diseases.
* Intake of medications on a regular basis, not including oral contraceptives for group 1 and 2.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2021-11-27 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
PCOS Rotterdam criteria | 3 months
  Ovary volume >9ml, presence of 12 or more follicles, biochemical or clinical signs of hyperandrogenism and anovulation.

SECONDARY OUTCOMES:
Insulin resistance (IR) | 3 months
  HOMA-IR was calculated with insulin and glucose fasting levels to determine the severity of insulin resistance

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Médico ABC, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided